CLINICAL TRIAL: NCT01270776
Title: Comparison of 2% Chlorhexidine in 70% Isopropyl Alcohol Versus 2% Aqueous Chlorhexidine for Skin Antisepsis Prior to Venepuncture in Very Low Birth Weight Infants: A Planned Non-inferiority Trial
Brief Title: Efficacy Study Comparing 2% Chlorhexidine in 70% Isopropyl Alcohol Versus 2% Aqueous Chlorhexidine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Vibhuti Shah, Staff Neonatologist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10 - 0112 - E
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Anti-infecting Agents, Local
Keywords: Randomized Controlled Trial; Chlorhexidine; Infant, Premature
MeSH Terms: conditions — Premature Birth | interventions — Chlorhexidine; 2-Propanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aqueous Chlorhexidine (Experimental): The group received skin antisepsis using 2% aqueous chlorhexidine solution.
  Interventions: Drug: 2% aqueous chlorhexidine
- 2% Chlorhexidine 70% isopropyl alcohol (Active Comparator): The group will receive skin antisepsis with 2% chlorhexidine solution in alcohol.
  Interventions: Drug: 2% Chlorhexidine 70% isopropyl alcohol

INTERVENTIONS:
Drug: 2% aqueous chlorhexidine — A single application of a swabstick impregnated with the antiseptic solution over the desired area. The imparted solution will be allowed to air dry with a minimum time of 30 seconds before intervention.
  Other Names: SOLU-I.V. Aqueous Swabsticks
  Arms: Aqueous Chlorhexidine
Drug: 2% Chlorhexidine 70% isopropyl alcohol — single application of a swabstick impregnated with the antiseptic solution over the desired area. The imparted solution will be allowed to air dry with a minimum time of 30 seconds before intervention.
  Other Names: SOLU-I.V. Swabsticks
  Arms: 2% Chlorhexidine 70% isopropyl alcohol

SUMMARY:
The purpose of this study is to compare the efficacy of two different antiseptic solutions (2%chlorhexidine in 70% alcohol with 2% aqueous chlorhexidine)when used in a standardized controlled manner in cleansing the skin of infants with birth weight less than 1500 grams prior to a skin breaking procedure (venepuncture).

The investigators hypothesize that the use of limited amount of 2% aqueous chlorhexidine solution will be as effective as the same amount of 2% chlorhexidine in 70% alcohol for skin antisepsis and that limited exposure to 2% aqueous CHG may be associated with less adverse skin reactions.

Literature from adults has shown that both 2% chlorhexidine in 70% alcohol as well as 2% aqueous chlorhexidine can provide effective skin antisepsis though alcohol containing solution had more long lasting effect. It is also well known from many case reports that alcohol containing products when used to clean abdominal skin for neonatal procedures can cause severe skin damage in preterm infants. This has lead many neonatal units to adopt aqueous chlorhexidine as the antiseptic agent of choice without robust evidence to support its use or standardization of method of application.Both these solutions are widely used in neonatal intensive care units across the globe including Canada.

By conducting this trial, the investigators want to evaluate the efficacy and safety of 2% aqueous chlorhexidine as an antiseptic agent when used in a controlled manner [limited amount for short duration].

DETAILED DESCRIPTION:
Venepuncture, either to obtain blood samples for laboratory investigations or to place peripheral intravascular catheters, is an integral part of care in neonatal intensive care units (NICUs). In sick neonates, apart for collection of blood samples venous cannulation is necessary for provision of total parenteral nutrition and administration of medications; however, these skin-breaking procedures places them at risk for local and systemic infectious complications. Bacterial organisms inhabited on the skin travel through the insertion site into the catheter tract and colonize the catheter tip. This is postulated to be a common route of infection for peripherally inserted catheters, hence the need for maintaining optimal skin antisepsis during such procedures.

It is not possible to completely sterilize the skin; however skin antisepsis aims to reduce the number of viable resident organisms on or in the skin and to destroy pathogenic organisms that may be on the skin. Several antiseptic agents are available for skin preparation including 70% alcohol, chlorhexidine (with 70% alcohol or aqueous) and povidone-iodine (PI). Most of the studies comparing the efficacy to these agents have been conducted in adults while there is paucity of studies regarding their use in VLBW infants.

Chlorhexidine, one of the most commonly used biocide antiseptic product, is a broad spectrum bactericidal agent. It diffuses through the outer cell wall and then attacks the bacterial cytoplasmic or inner membrane leading to cell death. Chlorhexidine is active against common gram negative and gram positive pathogens as well as yeast. Numerous randomized controlled trials have been performed in adult patients supporting the superiority of chlorhexidine as skin disinfectant. One of the more influential studies was conducted by Hibbard et al in 2002. The investigators compared 70% isopropyl alcohol; 2% CHG in 70% alcohol; and 2% aqueous CHG in healthy volunteers by obtaining abdominal and inguinal skin swabs at various time points after application. They concluded that all three solutions had excellent and comparable immediate antimicrobial action at 10 minutes & 6 hours after application but 2% CHG in 70% alcohol had better persistent action with antisepsis effectiveness at 24 hours. To date, this is the only study that has compared 2% CHG with and without alcohol directly.

Even though all the above mentioned solutions have proven excellent safety profile in adults, there are significant concerns with their use in preterm neonates. The skin of the newborn infant, especially the preterm infant, is more susceptible to damage from antiseptic agents. Iodine preparations have been associated with transient suppression of thyroid function related to systemic absorption. Alcohol and iodine have been reported to be associated with severe skin injury including blistering, burns and sloughing. Systemic absorption of chlorhexidine is rare, although it has been reported to occur when alcohol is used concurrently. These adverse events have only been reported when these solutions were used for placements of umbilical lines presumably because larger surface area of skin is exposed to a greater quantity of solution for longer duration. Also during such procedures the solution can often get pooled over abdominal skin if used in excessive quantity. No serious adverse event has ever been reported during venepuncture (from either form of chlorhexidine). Such significant concerns with the use of iodine and alcohol containing solutions and more widespread availability of aqueous chlorhexidine has led many NICU's to endorse its use without systematically evaluating its efficacy in this population or standardization of method of application. Therefore, it is important to conduct a well designed study to systematically evaluate the effectiveness of using a limited amount of 2% aqueous CHG in clinical practice.

This double blind planned non-inferiority randomized controlled trial will compare the efficacy and safety of 2% chlorhexidine in 70% isopropyl alcohol (current standard of practice in the NICU) to 2% aqueous chlorhexidine (investigational agent) for skin antisepsis prior to venepuncture in very low birth weight (VLBW, birth weight < 1,500 grams) infants. The effectiveness (success) of skin antisepsis will be assessed by collecting pre- and post- cleansing skin swabs. The skin swabs will then be cultured in the microbiology laboratory and pre- and post- microbial growth will be compared between the two groups.

Changes to the study protocol:

1. Results of the interim analysis:

   Following the pre-planned interim analysis, it is shown that the initial assumption of standard solution clearance rate used for sample size calculation (92%) was higher than the rate actually observed in the dataset collected up to the interim analysis stage by the investigators (84%). With the assumption of 84% clearance rate for standard solution, the study would have required a bigger sample size of 231 subjects in each arm. With the interim data, the two groups show exactly the same rates of clearance (84%) but with wide confidence intervals for the clearance rate estimates due to smaller sample size. Based on this interim analysis we do not statistically show non-inferiority of the test solution to standard solution. However to obtain a definitive answer we now need to modify our sample size to 462 subjects (231 subjects per arm).
2. This will now be a multi-center study. We have added SickKids, Toronto as an additional site for recruitment. We have obtained REB approval from SickKids.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1500 grams
* Postnatal age > 48 hours and < 28 days
* Need for venepuncture for any medical indication

Exclusion Criteria:

* Birth weight ≥ 1500 grams
* Infants with skin breakdown or previously documented to have skin reactions to antiseptic agent

Ages: 48 Hours to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 462 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial colony count as assessed by pre- and post cleansing skin swab culture. | 24 hours
  A sterile cotton swab with be rolled 4 times across the sampling area. The swab will be broken off into tube containing 1ml of sterile normal saline. A 0.1ml aliquot of this solution will be spread onto a blood agar plate. Colony forming units (CFU) will be enumerated after aerobic incubation at 37°C for 24 hours. Swabs which yield CFU > 15 will be labeled positive for bacteria and negative if CFU < 15.

SECONDARY OUTCOMES:
Immediate or late Skin reactions. | 24 hours
  Local adverse events will be recorded by researcher at 10 minutes after the procedure and then again at 2, 12 and 24 hours later to monitor for immediate and late local reactions. Adverse events will be recorded using a validated contact dermatitis score.

CONTACTS AND LOCATIONS:
Overall Officials: Vibhuti Shah, MD MRCP, Study Chair — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Keyworth N, Millar MR, Holland KT. Development of cutaneous microflora in premature neonates. Arch Dis Child. 1992 Jul;67(7 Spec No):797-801. doi: 10.1136/adc.67.7_spec_no.797. PMID 1519978
- [Background] D'Angio CT, McGowan KL, Baumgart S, St Geme J, Harris MC. Surface colonization with coagulase-negative staphylococci in premature neonates. J Pediatr. 1989 Jun;114(6):1029-34. doi: 10.1016/s0022-3476(89)80457-3. PMID 2723895
- [Background] McDonnell G, Russell AD. Antiseptics and disinfectants: activity, action, and resistance. Clin Microbiol Rev. 1999 Jan;12(1):147-79. doi: 10.1128/CMR.12.1.147. PMID 9880479
- [Background] Maki DG, Ringer M, Alvarado CJ. Prospective randomised trial of povidone-iodine, alcohol, and chlorhexidine for prevention of infection associated with central venous and arterial catheters. Lancet. 1991 Aug 10;338(8763):339-43. doi: 10.1016/0140-6736(91)90479-9. PMID 1677698
- [Background] Chaiyakunapruk N, Veenstra DL, Lipsky BA, Saint S. Chlorhexidine compared with povidone-iodine solution for vascular catheter-site care: a meta-analysis. Ann Intern Med. 2002 Jun 4;136(11):792-801. doi: 10.7326/0003-4819-136-11-200206040-00007. PMID 12044127
- [Background] Valles J, Fernandez I, Alcaraz D, Chacon E, Cazorla A, Canals M, Mariscal D, Fontanals D, Moron A. Prospective randomized trial of 3 antiseptic solutions for prevention of catheter colonization in an intensive care unit for adult patients. Infect Control Hosp Epidemiol. 2008 Sep;29(9):847-53. doi: 10.1086/590259. PMID 18665819
- [Background] Hibbard JS, Mulberry GK, Brady AR. A clinical study comparing the skin antisepsis and safety of ChloraPrep, 70% isopropyl alcohol, and 2% aqueous chlorhexidine. J Infus Nurs. 2002 Jul-Aug;25(4):244-9. doi: 10.1097/00129804-200207000-00007. PMID 12131506
- [Background] Malathi I, Millar MR, Leeming JP, Hedges A, Marlow N. Skin disinfection in preterm infants. Arch Dis Child. 1993 Sep;69(3 Spec No):312-6. doi: 10.1136/adc.69.3_spec_no.312. PMID 8215573
- [Background] Garland JS, Buck RK, Maloney P, Durkin DM, Toth-Lloyd S, Duffy M, Szocik P, McAuliffe TL, Goldmann D. Comparison of 10% povidone-iodine and 0.5% chlorhexidine gluconate for the prevention of peripheral intravenous catheter colonization in neonates: a prospective trial. Pediatr Infect Dis J. 1995 Jun;14(6):510-6. doi: 10.1097/00006454-199506000-00008. PMID 7667056
- [Background] Baumgartner C, Constant H, Putet G, Aulagner G. Cutaneous antiseptic efficacy of two ethanol chlorhexidine dilutions for neonatal venepuncture. Journal De Pharmacie Clinique 1998;17:109-12.
- [Background] Linder N, Prince S, Barzilai A, Keller N, Klinger G, Shalit I, Prince T, Sirota L. Disinfection with 10% povidone-iodine versus 0.5% chlorhexidine gluconate in 70% isopropanol in the neonatal intensive care unit. Acta Paediatr. 2004 Feb;93(2):205-10. doi: 10.1080/08035250310008159. PMID 15046275
- [Background] Lilley C, Powls A, Gray A. A prospective randomised double blind Comparison of 0.5% versus 0.05% aqueous Chlorhexidine for skin antisepsis prior to line insertion in neonates. Arch. Dis. Child. 2006;91;17-19.
- [Background] Garland JS, Alex CP, Uhing MR, Peterside IE, Rentz A, Harris MC. Pilot trial to compare tolerance of chlorhexidine gluconate to povidone-iodine antisepsis for central venous catheter placement in neonates. J Perinatol. 2009 Dec;29(12):808-13. doi: 10.1038/jp.2009.161. Epub 2009 Oct 8. PMID 19812587
- [Background] Mannan K, Chow P, Lissauer T, Godambe S. Mistaken identity of skin cleansing solution leading to extensive chemical burns in an extremely preterm infant. Acta Paediatr. 2007 Oct;96(10):1536-7. doi: 10.1111/j.1651-2227.2007.00376.x. Epub 2007 Aug 28. PMID 17727692
- [Background] Reynolds PR, Banerjee S, Meek JH. Alcohol burns in extremely low birthweight infants: still occurring. Arch Dis Child Fetal Neonatal Ed. 2005 Jan;90(1):F10. doi: 10.1136/adc.2004.054338. No abstract available. PMID 15613563
- [Background] Upadhyayula S, Kambalapalli M, Harrison CJ. Safety of anti-infective agents for skin preparation in premature infants. Arch Dis Child. 2007 Jul;92(7):646-7. doi: 10.1136/adc.2007.117002. No abstract available. PMID 17588981
- [Background] Datta MK, Clarke P. Current practices in skin antisepsis for central venous catheterisation in UK tertiary-level neonatal units. Arch Dis Child Fetal Neonatal Ed. 2008 Jul;93(4):F328. doi: 10.1136/adc.2008.137430. No abstract available. PMID 18567744
- [Background] Keyworth N, Millar MR, Holland KT. Swab-wash method for quantitation of cutaneous microflora. J Clin Microbiol. 1990 May;28(5):941-3. doi: 10.1128/jcm.28.5.941-943.1990. PMID 2191014
- [Background] Maki DG, Ringer M. Evaluation of dressing regimens for prevention of infection with peripheral intravenous catheters. Gauze, a transparent polyurethane dressing, and an iodophor-transparent dressing. JAMA. 1987 Nov 6;258(17):2396-403. PMID 3118061
- [Derived] Jain A, Deshpande P, Yoon EW, Lee KS, McGeer A, Shah V. 2% aqueous vs alcohol-based chlorhexidine for skin antisepsis in VLBW neonates undergoing peripheral venipuncture: a non-inferiority trial. J Perinatol. 2022 May;42(5):636-641. doi: 10.1038/s41372-022-01337-1. Epub 2022 Feb 19. PMID 35184146